CLINICAL TRIAL: NCT03557359
Title: A Phase II, Open Label, Single Arm Study of Nivolumab for Recurrent or Progressive IDH Mutant Gliomas With Prior Exposure to Alkylating Agents
Brief Title: Nivolumab for Recurrent or Progressive IDH Mutant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fabio Iwamoto, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Fabio Iwamoto, MD, Assistant Professor of Neurology at the Columbia University Medical Center, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6354
Record Dates: First submitted 2018-05-17; First posted 2018-06-15 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Gliomas
Keywords: Recurrent; Progressive; High Grade Glioma; IDH Mutant; Low Grade Glioma
MeSH Terms: conditions — Glioma; Recurrence | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 240 mg will be given every 2 weeks for 8 cycles. Beginning with Cycle 9, nivolumab 480 mg will be given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab will be administered as a 30-minute infusion. A finite treatment duration with immune therapies in this participant population remains an area of ongoing research; therefore the treatment duration chosen was 2 years.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (Opdivo®) is a human monoclonal antibody (HuMAb; immunoglobulin G4 (IgG4)- S228P) that targets the PD-1 cluster of differentiation 279 (CD279) cell surface membrane receptor.
  Other Names: Opdivo®

SUMMARY:
The objective of this study is to determine response rates (partial and complete responses) to nivolumab of recurrent or progressive IDH mutant (grades 2, 3 or 4) gliomas with prior exposure to alkylating agents.

DETAILED DESCRIPTION:
Gliomas are the most common malignant primary brain tumor in adults. Their clinical presentation is heterogeneous and prognosis is dependent on both the grade of the tumor and the molecular subtype. Somatic mutations in Isocitrate dehydrogenase 1 (IDH1) or, less commonly, Isocitrate dehydrogenase 2 (IDH2) genes have emerged as an important prognostic factor in gliomas and are associated with longer survival.

Regardless of initial grade, recurrence and transformation into higher grade tumors is almost universal. There is high unmet medical need in treating recurrent gliomas as there is currently no established standard of care therapy. Recent trials of IDH inhibitors in IDH mutant gliomas and programmed cell death protein 1 (PD-1) and PD-L1 inhibitors in recurrent gliomas have been disappointing. Multiple studies in other cancers have demonstrated that hypermutated tumors are associated with response to immunotherapeutic agents, including anti-CTLA4 agents in melanoma, anti-PD1 therapy in bladder cancer, and anti-programmed-cell-death protein 1 (anti-PD1) therapy in lung, and colorectal cancer.

There is evidence to suggest that gliomas with somatic IDH mutations are more prone to develop hypermutation after exposure to alkylating agents than IDH wildtype tumors, providing strong scientific rationale for establishing nivolumab as a treatment option in this subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.
* Participant must be 18 years of age or older
* Participants with pathologically confirmed grade 2, 3 or 4 gliomas with IDH mutation (confirmed by IDH R132H immunohistochemistry or IDH1/IDH2 next generation sequencing) who have progressive tumor and have had previous exposure to alkylating agents.
* Participants must have measurable disease, defined as at least one enhancing tumor lesion that can be accurately measured in at least one dimension as ≥ 10mm x 10mm on brain MRI. See 13.2 Disease Parameters for more information regarding evaluation of measurable disease. Patients with non-enhancing measureable disease may be eligible upon discussion with and approval by the CUMC PI.
* Availability of baseline frozen tumor or formalin-fixed paraffin-embedded (FFPE) tumor block.
* Karnofsky Performance Score (KPS) of 60 and above
* Adequate bone marrow, kidney and liver function as defined below:

  i) White blood count (WBC) ≥ 3000/microliter (uL) ii) Neutrophils ≥ 1500/uL iii) Absolute lymphocyte count ≥ 500/uL iv) Platelets ≥ 100x103 /uL v) Hemoglobin ≥ 9.0g/dL vi) Serum creatinine ≤ 1.5x upper limit of normal (ULN) or calculated creatinine clearance (CrCl)> 50 mL/min (using the Cockcroft-Gault formula)
  1. Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  2. Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL vi) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN vii) Total bilirubin (TBILI) ≤ 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0xULN)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study drug
* Women must not be pregnant or breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 5 months after the last dose of study treatment (i.e., 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives.)
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment (i.e., 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five halflives.)
* Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but still must undergo pregnancy testing.
* Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly.
* At a minimum, participants must agree to use 1 highly effective method of contraception

Exclusion Criteria:

* Participants with an active, known, or suspected autoimmune disease.
* Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Dose of dexamethasone ≤ 4 mg/day or equivalent is allowed at the study entry for brain tumor edema
* Participants who have received chemotherapy or experimental agents within 4 weeks (except for 6 weeks for nitrosoureas and 23 days for temozolomide) and radiotherapy within 12 weeks of the first dose of the study treatment.
* Prior use of PD-1, PD-L1, or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors or exposure to other checkpoint inhibitors.
* Prior exposure to bevacizumab or other vascular endothelial growth factor (VEGF) or VEGFR inhibitors.
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection, and/or detectable virus
* History of severe allergy or hypersensitivity to nivolumab components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2025-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Iwamoto, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Miami Cancer Center, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan H, Parsons DW, Jin G, McLendon R, Rasheed BA, Yuan W, Kos I, Batinic-Haberle I, Jones S, Riggins GJ, Friedman H, Friedman A, Reardon D, Herndon J, Kinzler KW, Velculescu VE, Vogelstein B, Bigner DD. IDH1 and IDH2 mutations in gliomas. N Engl J Med. 2009 Feb 19;360(8):765-73. doi: 10.1056/NEJMoa0808710. PMID 19228619
- [Background] Kirkpatrick JP, Sampson JH. Recurrent malignant gliomas. Semin Radiat Oncol. 2014 Oct;24(4):289-98. doi: 10.1016/j.semradonc.2014.06.006. PMID 25219814
- [Background] Burris H MI, Maher E, et al. Abstract PL04-05: The first reported results of AG-120, a first-in-class, potent inhibotior of the IDH1 mutant protein, in a Phase I study of patients with advanced IDH1-mutant solid tumors, including gliomas. Molecular Cancer Therapeutics 2015;14.
- [Background] Sampson JH OA, Vlahovic G, Sahebjam S, Baehring J, Hafler D, Voloschin A, Latek R, Cloughesy T, Lim M, Reardon D. Safety and Activity of Nivolumab +/- Ipilimumab in Recurrent Glioblastoma: Updated Results from CHECKMATE-143. Journal of Neurosurgery 2016;124:A1189-A90.
- [Background] Campesato LF, Barroso-Sousa R, Jimenez L, Correa BR, Sabbaga J, Hoff PM, Reis LF, Galante PA, Camargo AA. Comprehensive cancer-gene panels can be used to estimate mutational load and predict clinical benefit to PD-1 blockade in clinical practice. Oncotarget. 2015 Oct 27;6(33):34221-7. doi: 10.18632/oncotarget.5950. PMID 26439694
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] LeBlanc VG, Marra MA. Next-Generation Sequencing Approaches in Cancer: Where Have They Brought Us and Where Will They Take Us? Cancers (Basel). 2015 Sep 23;7(3):1925-58. doi: 10.3390/cancers7030869. PMID 26404381
- [Background] Cahill DP, Levine KK, Betensky RA, Codd PJ, Romany CA, Reavie LB, Batchelor TT, Futreal PA, Stratton MR, Curry WT, Iafrate AJ, Louis DN. Loss of the mismatch repair protein MSH6 in human glioblastomas is associated with tumor progression during temozolomide treatment. Clin Cancer Res. 2007 Apr 1;13(7):2038-45. doi: 10.1158/1078-0432.CCR-06-2149. PMID 17404084

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-five patients were enrolled and 33 patients received at least one dose of nivolumab. Two patients were lost to follow up before beginning treatment. Thirty-two patients completed the full 2-year treatment and one patient discontinued after 23 months due to Grade 2 transaminitis. Thirty-three patients were included in the analysis.
Groups:
- Nivolumab 240 mg: Nivolumab 240 mg will be given every 2 weeks for 8 cycles. Nivolumab will be administered as a 30-minute infusion. A finite treatment duration with immune therapies in this participant population remains an area of ongoing research; therefore the treatment duration chosen was 2 years.
  Nivolumab: Nivolumab (Opdivo®) is a human monoclonal antibody (HuMAb; immunoglobulin G4 (IgG4)- S228P) that targets the PD-1 cluster of differentiation 279 (CD279) cell surface membrane receptor.
- Nivolumab 480 mg: Beginning with Cycle 9, Nivolumab 480 mg will be given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent. Nivolumab will be administered as a 30-minute infusion. A finite treatment duration with immune therapies in this participant population remains an area of ongoing research; therefore the treatment duration chosen was 2 years.
  Nivolumab: Nivolumab (Opdivo®) is a human monoclonal antibody (HuMAb; immunoglobulin G4 (IgG4)- S228P) that targets the PD-1 cluster of differentiation 279 (CD279) cell surface membrane receptor.
Period: Dose 1: 240 mg
Arm/Group | Nivolumab 240 mg | Nivolumab 480 mg
Started | 33 | 0
Completed | 32 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Dose 2: 480 mg
Arm/Group | Nivolumab 240 mg | Nivolumab 480 mg
Started | 0 | 13
Completed | 0 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 44.5 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 35
Recurrent or progressive IDH mutant (grades 2, 3 or 4) gliomas in subjects 18 years of age or older [Count of Participants; unit: Participants] | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The overall response rate is defined as the percentage of patients with a reduction in tumor size while on treatment.
Time Frame: Throughout treatment duration or until progressive disease, unacceptable toxicity, or withdrawal of consent, up to 2 years
Measure: Number; unit: percent
Arm/Group | Nivolumab
Number analyzed (Participants) | 33
percent | 9

2. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Until the first date that progressive disease is objectively documented or until study completion (36 months)
Reporting Status: Not Posted

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Participants discontinuing study treatment will remain on study for documentation of progression and death.
Time Frame: Until death or study completion (36 months)
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of nivolumab to death due to any cause. All other participants will be censored at the last date known to be alive.
Time Frame: Until death or study completion (36 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- Nivolumab 240 mg: Nivolumab 240 mg will be given every 2 weeks for 8 cycles.
- Nivolumab 480 mg: Beginning with Cycle 9, Nivolumab 480 mg will be given every 4 weeks for a total therapy duration of 2 years, or until progressive disease, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Nivolumab 240 mg | Nivolumab 480 mg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/13
Serious Adverse Events (participants affected / at risk) | 9/33 | 4/13
Other Adverse Events (participants affected / at risk) | 29/33 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 240 mg (N=33) | Nivolumab 480 mg (N=13)
Hypotension (Vascular disorders) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Muscle weakness - Right Side (Musculoskeletal and connective tissue disorders) | 1 | 1
Stroke (Nervous system disorders) | 0 | 2
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Muscle weakness - Left Side (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nivolumab 240 mg (N=33) | Nivolumab 480 mg (N=13)
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1
Allergic reaction (Immune system disorders) | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3
Autoimmune disorder (Immune system disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 2
Dizziness (Nervous system disorders) | 4 | 2/12
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dysphasia (Nervous system disorders) | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Edema limbs (General disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Facial muscle weakness (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3
Fatigue (General disorders) | 9 | 3
Flashing lights (Eye disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 3
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Lethargy (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 6 | 2
Memory impairment (Nervous system disorders) | 2 | 1
Mucosal infection (Infections and infestations) | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 4 | 1
Neutrophil count decreased (Infections and infestations) | 1 | 0
Pain (General disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Reproductive system and breast disorders) | 1 | 2
Restlessness (Psychiatric disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 3
Serum amylase increased (Investigations) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 3
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Weight gain (Investigations) | 1 | 1
Weight loss (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03557359/Prot_SAP_000.pdf